CLINICAL TRIAL: NCT00993837
Title: Comparison of Effectiveness and Safety of Thyroidectomy for Thyroid Carcinoma in Patients Undergo Endoscopic Surgery and Those Receive Conversion
Brief Title: Feasibility of Endoscopic Thyroidectomy for Thyroid Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Military Medical University (Other)
Responsible Party: Minimally Invasive Surgical Center, Changzheng Hospital, Second Military Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SMMU-2-2009-3
Record Dates: First submitted 2009-09-29; First posted 2009-10-14 (Estimated); Last update posted 2009-10-14 (Estimated); Status verified 2009-10

CONDITIONS: Thyroid Carcinoma
Keywords: endoscopic thyroidectomy; thyroid carcinoma
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Thyroidectomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- conversion (Experimental)
  Interventions: Procedure: thyroidectomy

INTERVENTIONS:
Procedure: thyroidectomy — total thyroidectomy via endoscopic approach and that convert to open procedure
  Other Names: totally endoscopic thyroidectomy

SUMMARY:
Endoscopic thyroidectomy has been used to treat thyroid diseases in China. However, whether this technique is rational to treat thyroid carcinoma is still in controversy. The diagnosis of thyroid carcinoma is predominantly made according to intra-operative frozen section pathological examination in China. In this research, the investigators want to compare clinical index (blood loss, operation duration, number of lymph nodes dissected, complication rates, etc) between patients underwent endoscopic thyroidectomy ( total thyroidectomy) and those underwent conversion to open procedure. The investigators want to evaluate the technical feasibility of endoscopic thyroidectomy for treating thyroid carcinoma.

DETAILED DESCRIPTION:
intra-operative diagnosis of thyroid carcinoma is usually considered the indication of conversion to open surgery. with accumulation of experience of endoscopic thyroidectomy, the investigators want to evaluate the technical feasibility, completeness and safety of endoscopic thyroidectomy.

ELIGIBILITY:
Inclusion Criteria:

* lesion diameter less than 1 cm by ultrasound

Exclusion Criteria:

* frozen section diagnosis indicates benign lesion

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-12 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
to evaluate the completeness of thyroid resection and clearance of lymph nodes in the central compartment, and to observe the complications such as RLN palsy and hypocalcemia | 1 year after operation

CONTACTS AND LOCATIONS:
Overall Officials: Ming QIU, Dr., Study Chair — Changzheng Hospital affliated to SMMU
Locations (1):
- Changzheng Hospital, Shanghai, Shanghai Municipality, China